CLINICAL TRIAL: NCT00820326
Title: A Randomized, Double-Blind, Placebo-Controlled, Study of Efficacy of DOLASETRON in Patients With Fibromyalgia
Brief Title: Efficacy of Dolasetron in Patients With Fibromyalgia
Acronym: Dolastron
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Limoges (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: I03002
Record Dates: First submitted 2008-12-27; First posted 2009-01-12 (Estimated); Last update posted 2025-07-16 (Actual); Status verified 2009-01

CONDITIONS: Fibromyalgia
MeSH Terms: conditions — Fibromyalgia | interventions — dolasetron

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dolasetron (Active Comparator): Patients will receive dolasetron at a dose of 12.5 mg / day for 4 days at J0, M1, M2 and M3
  Interventions: Drug: Dolasetron
- Placebo (Placebo Comparator): Patients will receive placebo everyday for 4 days at J0, M1, M2 and M3
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dolasetron — Patients will receive dolasetron at a dose of 12.5 mg / day for 4 days at J0, M1, M2 and M3
  Arms: Dolasetron
Drug: Placebo — Patients will receive placebo everyday for 4 days at J0, M1, M2 and M3
  Arms: Placebo

SUMMARY:
This study offers a new treatment, dolasetron or ANZEMET ®, which will be administered by intravenous way once a day during a 4 days Hospitalization.

This study is double blind (neither you nor the physician will know if you are receiving active study drug or placebo).

Randomisation at the beginning of the study will decide whether you receive active treatment or its placebo.

This treatment will be renewed after one month, after 2 months and after 3 months.

If the study staff determines that you are eligible and you decide to participate, there will be approximately 6 study visits in about 9 months. During these visits, you will undergo routine health exams and complete different kinds of questionnaires.

Following this first period of 3 months, you agree to come back for consultation at month 4, month 6 and month 12 for monitoring and evaluating the effects of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 to 75
* Primitive Fibromyalgia according to ACR criteria
* Patient no responding to conventional treatment
* Women of childbearing age using an efficace contraception
* Signed consent

Exclusion Criteria:

* Inflammatory rheumatic diseases
* Diseases of the system: Gougerot Sjögren, polymyositis, vasculitis,
* Infectious diseases: hepatitis B and C, lyme disease, HIV,
* Hypothyroidism,
* Bone and mineral metabolism disorders
* Disorders of cardiac conduction
* Failure of Heart, of kidney or liver,
* Patient allergic to dolasetron
* Pregnant or nursing women
* Women without means of contraception,
* Age <18 or > 75 years.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2004-03; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Measure: Improving visual analogue scale (VAS) between Inclusion visit and month 3 | Inclusion visit and month 3

SECONDARY OUTCOMES:
Improving visual analogue scale (VAS) | Between Inclusion visit, month 1, month 2, month 4, month 6, and month 12.
Fibromyalgia impact questionnaire SF-36 scale and Beck depression scale | Between Inclusion visit, month 1, month 2, month 4, month 6, and month 12.
Anxiety index | Between Inclusion visit, month 1, month 2, month 4, month 6, and month 12.
Number of painful trigger points | Between Inclusion visit, month 1, month 2, month 4, month 6, and month 12.

CONTACTS AND LOCATIONS:
Locations (1):
- Service de Rhumatologie, CHu de Limoges, Limoges, France

REFERENCES:
- [Result] Vergne-Salle P, Dufauret-Lombard C, Bonnet C, Simon A, Treves R, Bonnabau H, Bertin P. A randomised, double-blind, placebo-controlled trial of dolasetron, a 5-hydroxytryptamine 3 receptor antagonist, in patients with fibromyalgia. Eur J Pain. 2011 May;15(5):509-14. doi: 10.1016/j.ejpain.2010.09.013. Epub 2010 Oct 30. PMID 21036635